CLINICAL TRIAL: NCT01864044
Title: Prospective Observational Lymphoedema Intensive Treatment
Acronym: POLIT
Status: Completed | Type: Observational
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Other Study IDs: EC07
Record Dates: First submitted 2013-05-13; First posted 2013-05-29 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Lymphoedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of this observational study was to describe usual practices in lymphedema management in France.

It was the opportunity to assess the effects of these practices on lymphedema volume in a large number of patients, to identify predictive factors of response, and to assess the safety of this therapy.

DETAILED DESCRIPTION:
Lymphoedema is commonly treated according a strategy called Complex Decongestive Therapy (CDT). This CDT is usually composed of 2 different treatment phases. The first phase is an acute phase which aim is to reduce affected limb volume. The second phase is a maintenance phase which aim is to maintain as long as possible the volume reduction acheived during the first phase.

These 2 phases required multi modal parameters such as bandages, lymphatic drainages, physical exercises...and can be managed very differently from one site to another.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult patients
* hospitalized with a clinical diagnosis of unilateral stage II-III upper or lower limb lymphoedema of any etiology
* indication for intensive decongestive therapy (IDT)

Exclusion Criteria:

* bilateral lymphedema,
* lymphedema of both upper and lower limbs,
* intensive decongestive therapy in the previous 6 months,
* cancer recurrence,
* systolic pressure index < 0.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients hospitalized with a clinical diagnosis of unilateral stage II-III upper or lower limb lymphoedema of any etiology and an indication for intensive decongestive therapy (IDT) were enrolled.
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in affected limb volume | At the end of 1st phase of Complex Decongestive Therapy and 6 months later
  According to the site, the first phase can lasts 1, 2 or 3 weeks.